CLINICAL TRIAL: NCT07115719
Title: Early Decision Effect of Withholding and/or Withdrawing Life-sustaining Treatment on Emergency Department Patients' Short- and Long-term Outcomes: a Retrospective Analysis.
Brief Title: Withholding and/or Withdrawing Life-sustaining Treatment on Emergency Department Patients' Short- and Long-term Outcomes
Status: Completed | Type: Observational
Sponsor: Beaujon Hospital (Other)
Responsible Party: Principal Investigator, Prabakar VAITTINADA AYAR, doctor, Beaujon Hospital
Other Study IDs: urgBjNWHWD
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: WITHOLDING WITHDRAWING in End of Life Situation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — NO INTERVENTION

SUMMARY:
Background In France, a significant proportion of end-of-life (EOL) decisions occur in emergency departments (EDs), where time constraints and limited resources may hinder optimal care. Although withholding or withdrawing life-sustaining treatments (WHWD) is common in this context, the impact of timing on patient outcomes remains unclear.

Objective:

To assess how the timing of WHWD decisions influences short- and long-term outcomes among ED patients.

Methods:

We conducted a retrospective, observational study at Beaujon Hospital's ED (Paris, France) between January 2020 and December 2021. We included 354 adult patients admitted to the observation unit with a WHWD decision. Patients were categorized into early (eWHWD) and late (lWHWD) groups based on the median time to decision. The primary endpoint was 28-day all-cause mortality. Cox regression was used for survival analysis, adjusting for age, sex, comorbidities, functional status, and severity of illness.

ELIGIBILITY:
Inclusion Criteria:

* To be included, patients hospitalised after their ED visit must be admitted to the observation unit (OU) in association with a mention of a withholding/withdrawing of the life-sustaining treatment in the ED medical record.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients in end of life situation with withholding or withdrawing decision
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | 28-days

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Beaujon, Clichy, Île-de-France (Paris), France

IPD SHARING:
Plan to Share IPD: No